CLINICAL TRIAL: NCT04967131
Title: The Immediate Effect of Proprioceptive Neuromuscular Facilitation on Pain and Maximal Mouth Opening in Temporomandibular Dysfunction: Pilot Study
Brief Title: Proprioceptive Neuromuscular Facilitation Exercises in Temporomandibular Dysfunction
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, Gizem Ergezen, Istanbul Medipol University Hospital
Other Study IDs: 10840098-604.01.01-E.60748
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Disorders; Pain
Keywords: Orofacial Pain; Proprioceptive Neuromuscular Facilitation; Therapeutic Management; Threshold Pressure; Temporomandibular Joint Disorders; Pressure Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain; Facial Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PNF group: Proprioceptive Neuromuscular Fascilitation exercises were given this group
  Interventions: Other: PNF exercises

INTERVENTIONS:
Other: PNF exercises — PNF exercises were applied in 3 sets of 15 repetitions based on movement in the diagonal plane, using head, neck and chin patterns. Contractions were sustained for at least 10 seconds.

SUMMARY:
Individuals who were diagnosed with reduction disc displacement by Research Diagnostic criteria for Temporomandibular Disorder (TMD / RDC) were included in the study. Proprioceptive neuromuscular facilitation exercises were performed for 30 minutes using neck jaw and tongue patterns with rhythmic stabilization (RS) and combination of isotonics (CI) techniques by physiotherapist. Maximal mouth openings were measured with caliper, pain intensities were measured with visual analogue scale and pressure pain thresholds with hand algometer.

DETAILED DESCRIPTION:
TMD patients who are diagnosed by TMD/RDC are firstly assessed by physiotherapist for maximal mouth opening(MMO), pain intensity and pressure pain threshold. Then they will taught exercises with rhythmic initiation which includes repetation of the patern and 15 repetitions are applied as warm-up period. Proprioceptive neuromuscular facilitation (PNF) exercises are performed in the neck and jaw patterns with rhythmic stabilization (RS) and combination of isotonics (CI) techniques. In the neck, right rotation-right lateral flexion, left rotation-left lateral flexion pattern, and the opening and closing pattern according to the working mechanics of the masseter and temporal muscle in the chin, RS and CI techniques are used. By providing maximum resistance in accordance with the needs of each individual, the RS protocol consist of isometric contractions that would not involve changing movements for 10 seconds. The combination of isotonics technique include combined concentric, isometric, and eccentric contraction of the agonist muscle for 5 seconds of each contraction without rest. CI exercises consist of 15 repetitions per set. A 30-second rest given between sets to include recovery. After exercises immediate MMO, pain intensity and pain treshold assessment will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 18-25 years female, admitted to the study with clenching, grinding, clicking, jaw pain when eating hard foods, and limited and painful mouth movements.

Exclusion Criteria:

* Having orthopedic, neurological or rheumatological cervical disorders which affect the jaw motions; receiving occlusal therapy as a companion to treatment, those who have an operation in the area of jaw, head and neck and those with vertigo that prevents head movements during exercises.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female were included in this study, since it is included in the literature that temporomandibular dysfunction is observed 4-6 times more frequently in women than men
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Treshold | the immediate effect will be measured as soon as the exercise is finished
  The pain threshold will be measured with an algometer at certain points on the muscles in the area where the exercise is applied.
Pain intensity | the immediate effect will be measured as soon as the exercise is finished
  The level of pain felt will be marked with a visual analog scale on a 10-centimeter paper.
Maximum mouth opening | the immediate effect will be measured as soon as the exercise is finished
  Individuals will be asked to open their mouths as much as they can, and mouth opening will be measured with a caliper.

SECONDARY OUTCOMES:
Unassisted opening | the immediate effect will be measured as soon as the exercise is finished
  the individual is told to open their mouth and the gap is measured with a caliper.
maximum unassisted opening | the immediate effect will be measured as soon as the exercise is finished
  Without trying to increase the mouth opening with hand or any help, the individual actively opens mouth as much as they can and the opening is measured with a caliper.
maximum assisted opening | the immediate effect will be measured as soon as the exercise is finished
  It is measured with a caliper by asking individuals to open their mouths as much as they can and open more by helping with their hands at the last point.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Atılgan, PhD, Study Chair — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)